CLINICAL TRIAL: NCT01254097
Title: Feasibility Study of Probiotics in Primary Care
Brief Title: Probiotics in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, William Curry, Professor, Family and Community Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Probiotic-1
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Antibiotic Side Effect
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Placebo Comparator): Participants are provided in double blinded fashion, probiotic given to take with antibiotics prescribed by their provider.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Participants are provided in double blinded fashion, Look alike placebo given to take with antibiotics prescribed by their provider.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic capsule, 2 capsules twice daily
  Other Names: Florajen 3

SUMMARY:
Antibiotics are lifesaving medicines and generally safe, yet unwanted side effects are common. While destroying illness-causing 'bad' bacteria, antibiotics can upset the protective 'good' bacteria in the body. This research will test if taking a probiotic with prescribed antibiotics will decrease the chance of having bothersome antibiotic-associated side effects.

DETAILED DESCRIPTION:
Objectives Several studies have demonstrated that probiotics can be helpful in preventing antibiotic-associated diarrhoea in hospitalized patients. However, the extent to which probiotics may benefit healthy adults taking a course of antibiotics has not been investigated in primary care. Furthermore, patient willingness to take a probiotic supplement concomitantly with antibiotics has not been explored. We aimed to conduct an exploratory study using probiotics in adults requiring an acute course of antibiotic therapy.

Methods Patients prescribed antibiotics for treatment of acute infections in an outpatient family practice setting were randomized to receive either a probiotic or placebo concurrently. Patients completed adherence diaries and daily symptom checklists to assess gastrointestinal and vaginal (women) symptoms and collect information about adherence.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 - 79 years of age with infection requiring an oral antibiotic.
* Must be able to be contacted via telephone.

Exclusion criteria:

* pregnancy,
* breast-feeding,
* those receiving tube feeding,
* those with diarrhea as a current symptom of present illness, and pre-existing illnesses that contribute to diarrhea such as inflammatory bowel disease,
* irritable bowel syndrome, colitis or celiac disease.
* Those undergoing active cancer treatments with chemotherapeutic or radiation therapy,
* immunocompromised persons,
* history of cardiac valvular disease,
* those taking a laxative or stool softener on a daily basis, as well as
* persons treated with an antibiotic in the previous 60 days,
* new antibiotic prescription that exceeds a 10 day course, or regular use of a probiotic within the previous three weeks (including daily ingestion of yogurt).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Rate of antibiotic associated diarrhea | two weeks after start of antibiotics
  Groups will be compared based on rates of antibiotic associated diarrhea, symptoms developing in the two week window of when antibiotics are started.

SECONDARY OUTCOMES:
Participant knowledge of probiotics | At participant recruitment
  Assess current knowledge of probiotics of participants at the time of recruitment to study

CONTACTS AND LOCATIONS:
Overall Officials: William J Curry, MD, MS, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- M.S. Hershey Medical Center, Dept of Family and Community Medicine, Hershey, Pennsylvania, United States